CLINICAL TRIAL: NCT03005652
Title: A Multicenter Randomized Superiority Study To Compare The Effects Of An 8-Weeks Mindfulness-based Intervention Versus Health Education Programme On Mental Health And Wellbeing In Individuals With Subjective Cognitive Decline
Brief Title: Effects Of An 8-Weeks Mindfulness-based Intervention In Individuals With Subjective Cognitive Decline
Acronym: SCD-WELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: C16-61
Record Dates: First submitted 2016-12-16; First posted 2016-12-29 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Dysfunction
Keywords: Subjective Cognitive Decline; Mental Health; Meditation; Health Education
MeSH Terms: conditions — Cognitive Dysfunction; Psychological Well-Being; Health Education

STUDY DESIGN:
Intervention Model Description: The trial will compare outcomes in two groups of participants randomised to one of two study arms, either receiving:
  (i) an 8-week mindfulness-based intervention, using a secular form of mindfulness training; or (ii) an 8-week validated health-educational programme (comparison condition, see section 6.3 for description) The randomization will be performed with a 1:1 allocation. The primary outcome will be change in symptoms of anxiety from baseline to 8 weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness intervention (Experimental): consists of eight weekly group-based sessions of 2 hours duration and an individual pre-class interview, in which the participants will be socialised to the treatment. The intervention will combine intensive training in mindfulness and compassion meditation and gentle yoga practices with psycho-educational components targeted at helping individuals to deal more effectively with emotional difficulties and stressors commonly encountered in old age. These will include addressing concerns about cognitive functioning and health, and will have a particular emphasis on cultivating wholesome attitudes towards self and others.
  Interventions: Behavioral: Mindfulness weekly courses for 8 weeks
- Health education intervention (Active Comparator): follow the same format and structure as the mindfulness-based intervention, and will be matched to the mindfulness-based intervention in administration, dosage, and duration.
  The treatment is based on a published manual, with every session of the program covering different subjects, including self-management, problem-solving, sleep, stress, exercise, managing medicines and memory, communicating with family, friends, and healthcare professionals, eating, weight management, and planning for the future. Participants will be provided with information about these subjects and engage in group exercises and discussions about these subjects. They will be given a workbook and asked to actively engage in activities described in by the workbook to improve health and well-being on 6 out of 7 days each week, matching home assignments in the mindfulness-based intervention.
  Interventions: Behavioral: Health education weekly courses for 8 weeks

INTERVENTIONS:
Behavioral: Mindfulness weekly courses for 8 weeks — The mindfulness intervention combines intensive training in mindfulness and compassion meditations, light movement and yoga activities, and psycho-educational components to promote nonjudgmental awareness of present moment experiences.
  Arms: Mindfulness intervention
Behavioral: Health education weekly courses for 8 weeks — The health education intervention is group-based programme has been developed and validated in an SCD population. Each session of the course covers different subjects, which include self-management, problem-solving, sleep, stress, exercise, managing medicines and memory, communicating with healthcare professionals, eating, and planning for the future.
  Arms: Health education intervention

SUMMARY:
The European Commission Horizon 2020 programme has funded the SCD-WELL trial to investigate the efficacy of mindfulness-based training to reduce anxiety in individuals with Subjective Cognitive Decline (SCD), in comparison to an active comparison condition.

It is increasingly recognized that most neuropathological processes start years before the onset of clinical Alzheimer's disease (AD). Hence, there is a growing urgency to target individuals in the earliest stages for intervention when neurodegeneration is still limited. Individuals clinically judged to have SCD, defined by subjectively experienced cognitive decline but normal performance on cognitive tests, are at increased risk for future cognitive decline and AD. These individuals with SCD currently have no established treatment options. Symptoms of anxiety have high prevalence in this population, and evidence from recent longitudinal research links anxiety with significantly accelerated cognitive decline in at risk individuals. Effectively reducing anxiety in this population may therefore not only relieve participants from burdensome symptoms, but may also slow cognitive decline and delay or prevent the onset of AD.

The investigators chose to study the efficacy of a mindfulness-based intervention to reduce anxiety in this population because this type of intervention has been shown to reduce anxiety in a number of populations, including in older adults. Further, accumulating evidence indicates that intensive mindfulness training effectively down-regulates a number of other adverse psychological and biological risk factors for AD, such as stress, depression, insomnia, feelings of loneliness and social exclusion, and cardiovascular risk factors. These findings are relevant to AD because approximately a third of AD cases worldwide might be attributable to potentially modifiable risk factors. In spite of the increased use of mindfulness-based interventions to treat clinical symptoms, these trials often suffer from the lack of an adequate comparison condition and lack of follow up to know whether initial benefits are maintained.

DETAILED DESCRIPTION:
SCD-WELL includes both an active comparison condition and a 16-week follow up assessment after the end of the intervention. SCD-WELL is a non-CTIMP European multicentre, observer-blinded, randomized, controlled, superiority trial with two parallel groups, which compares anxiety and additional behavioural and biological outcomes amongst people with SCD who receive mindfulness-based training and those who receive a health education comparison intervention. Outcomes will be measured at baseline, post-intervention and 16 weeks after the end of the intervention.

160 older-adult patients diagnosed with SCD will be recruited to the study from memory clinics at four sites in Europe: London, UK; Cologne, Germany; Barcelona, Spain; Lyon, France where they will have sought help due to concern about their memory. Participants will be recruited in two waves over a maximum two-year period and will be provided with a participant information sheet, and asked to consider their participation. Should they wish to participate, and after a signed and dated Informed Consent Form has been obtained, a unique participant identification (ID) will be assigned to the participant.

Behavioural assessments will take place at baseline, after the intervention, and 16 weeks after the end of the intervention. Because we believe that mindfulness-based training has the potential to affect a number of areas of life we will also look at changes in other areas of psycho-affective symptoms, social functioning, awareness, well being and quality of life, sleep quality, and cognition, after the intervention and 16 weeks after the end of the intervention. Validated neuropsychological tests and behavioural questionnaires were selected for their sensitivity to the domains listed above. These measures will be completed alone by the participant or in the presence of a psychometrist. Questionnaires will also be completed by partners at the three time points to coincide with assessments of participants.

Blood samples will be taken at the memory clinic by certified phlebotomists at baseline, after the intervention and during follow-up to measure genetic markers of risk for AD as well as proteomic markers of stress and AD that may be affected by this intervention. Information will also be collected about the medical care of the participant.

Trained facilitators will deliver both interventions. Both interventions follow a manual, are group-based, include at-home activities, and are 8 weeks in duration. Both interventions provide individuals with sustainable skills that remain beyond the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 60 years
* Meet the research criteria proposed by the international SCD-I working group for studies in SCD
* Performance within the normal range on standardised cognitive tests according to agreed study-specific standards to rule out mild cognitive impairment (MCI) and dementia
* Either referred to the memory clinic by a physician or who are self-referrals because of memory concerns (assessed by a positive response to the question 'Are you worried about your memory?')
* Ability to provide informed consent in accordance with International Conference on Harmonization of Good Clinical Practice (GCP/ICH) guidelines and local regulations
* State that they are available for the trial duration

Exclusion Criteria:

* Presence of a major neurological or psychiatric disorder (including generalised anxiety, major depressive disorder, or an addiction to alcohol or drugs) according to ICD-10 and/or DSM 5 criteria
* Under legal guardianship or incapacitation
* History of cerebral disease (vascular, degenerative, physical malformation, tumor, or head trauma with loss of consciousness for more than an hour) which interferes with the aims of the study protocol
* Presence of a chronic disease or acute unstable illness (respiratory, cardiovascular, digestive, renal, metabolic, hematologic, endocrine or infectious) which interferes with the aims of the study protocol
* Current or recent medication that may interfere with cognitive action (psychotropic, systemic corticosteroid, anti-Parkinson's, or analgesic drugs). The interfering nature of the different treatments will be at the discretion of the investigating doctor.
* Have regularly or intensively practiced meditation or comparable practices (yoga, Qi Gong, Alexander technique)

  * more than one day per week for more than six months consecutively over the last 10 years,
  * intensively (internship or retreat > five consecutive days) over the past 10 years,
  * more than 25 days of retreats (cumulatively) prior to the last 10 years.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Mean change in anxiety after the intervention | Between baseline and the end of the 8-week interventions
  (measured by the trait-STAI)

SECONDARY OUTCOMES:
Mean change in anxiety from baseline to 24 weeks | From baseline and 24 weeks
  measured by the trait-STAI
Change in depression by the Geriatric Depression Scale (GDS) | a) from baseline to the end of the 8-week intervention b) from baseline to 24 weeks.
  depression (Geriatric Depression Scale) : Range 0-15, higher scores indicate greater depressive symptoms.
Change in behavioural measures of compassion measured by the Self Compassion and Compassionate Love Scale questionnaires | a) from baseline to the end of the 8-week intervention b) from baseline to 24 weeks.
  Self Compassion: Range 12-60, higher scores indicate greater compassion. Compassionate Love Scale: Range 21-147, higher scores indicate greater compassion.
Change in cognitive function assessed by a composite score derived from neuropsychological tests. | a) from baseline to the end of the 8-week intervention b) from baseline to 24 weeks.
  The composite score will correspond to the mean of z-scores calculated from relevant test scores from the Mattis Dementia Rating Scale-2 (DRS-2), Wechsler Adult Intelligence Scale-IV (WAIS-IV) Coding, Rey Auditory Verbal Learning Test (RAVLT), Category Fluency (Animals). Higher z-scores correspond to better cognitive performance.
Subjective measures of sleep collected via the Pittsburg Sleep Quality Index questionnaire | a) from baseline to the end of the 8-week intervention b) from baseline to 24 weeks.
  collected via the Pittsburg Sleep Quality Index questionnaire: Range 0-21, higher scores indicate better sleep quality
Change in lifestyle as assessed by The Physical Activity Scale for the Elderly questionnaire | a) from baseline to the end of the 8-week intervention b) from baseline to 24 weeks.
  assessed by The Physical Activity Scale for the Elderly questionnaire: Range 0-873, higher scores indicate more physical activity
Change in quality of life assessed by the world health organization quality of life - brief questionnaire | a) from baseline to the end of the 8-week intervention b) from baseline to 24 weeks.
  WHOQOL-bref: Range 21-147, higher scores indicate better quality of life.
Mean change in blood-based biological markers of stress and Alzheimer's disease assessed by DNA methylation patterns and quantities of proteins - neurofilament light and tau | a) from baseline to the end of the 8-week interventions and b) from baseline to 24 weeks.
  assessed by DNA methylation patterns and quantities of proteins - neurofilament light and tau

OTHER OUTCOMES:
Difference in partner perceptions of participant mindfulness measured by Five-Facet Mindfulness Questionnaire (FFMQ-15, range 15-75, higher scores indicate greater mindfulness) | a) from baseline to the end of the 8-week intervention and b) from baseline to 24 weeks.
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant.
Difference in partner perceptions of participant compassion towards others measured by Compassionate Love Scale (Range 21-147, higher scores indicate greater compassion) | a) from baseline to the end of the 8-week intervention and b) from baseline to 24 weeks.
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant.
Difference in partner perceptions of participant depression measured by the Geriatric Depression Scale (range 0-15, higher scores indicate greater depressive symptoms) | a) from baseline to the end of the 8-week intervention and b) from baseline to 24 weeks.
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant.
Difference in partner perceptions of participant anxiety measured by trait subscale of the state-trait anxiety inventory (trait-STAI, range 20-80, higher scores indicate greater anxiety symptoms) | a) from baseline to the end of the 8-week intervention and b) from baseline to 24 weeks.
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant.
Difference in partner perceptions of participant prosocialness measured by Prosocialness scale (range 16-80, higher scores indicate greater prosocialness) | a) from baseline to the end of the 8-week intervention and b) from baseline to 24 weeks.
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jessen, Principal Investigator — Director of the Clinic for Psychiatry and Psychotherapy at University Hospital Cologne; Natalie Marchant, Study Director — Division of Psychiatry, University College London
Locations (4):
- The Clinical Research Memory Centre of Lyon (CMRR), department of the University Hospitals of Lyon - Hospices Civils de Lyon (HCL), Lyon, France
- The Department of Psychiatry at University of Cologne (UKK), Cologne, Germany
- The Consorci Institut D'Investigacions Biomediques August Pi i Sunyer (IDIBAPS), Barcelona, Spain
- The Division of Psychiatry at University College London (UCL)., London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Masebo L, Whitfield T, Demnitz-King H, Heslegrave A, Poisnel G, Lutz A, Frison E, Wirth M, Hye A, Jessen F, Ashton NJ, Zetterberg H, Marchant NL. Can non-pharmacological interventions change levels of neurofilament light in older adults at risk of dementia? A secondary analysis of the SCD-Well randomized clinical trial. J Prev Alzheimers Dis. 2025 Sep;12(8):100299. doi: 10.1016/j.tjpad.2025.100299. Epub 2025 Jul 18. PMID 40683836
- [Result] D'elia Y, Whitfield T, Schlosser M, Lutz A, Barnhofer T, Chetelat G, Marchant NL, Gonneaud J, Klimecki O; Medit-Ageing group. Impact of mindfulness-based and health self-management interventions on mindfulness, self-compassion, and physical activity in older adults with subjective cognitive decline: A secondary analysis of the SCD-Well randomized controlled trial. Alzheimers Dement (Amst). 2024 Mar 4;16(1):e12558. doi: 10.1002/dad2.12558. eCollection 2024 Jan-Mar. PMID 38440222
- [Result] Marchant NL, Barnhofer T, Klimecki OM, Poisnel G, Lutz A, Arenaza-Urquijo E, Collette F, Wirth M, Schild AK, Coll-Padros N, Reyrolle L, Horney D, Krolak-Salmon P, Molinuevo JL, Walker Z, Maillard A, Frison E, Jessen F, Chetelat G; SCD-WELL Medit-Ageing Research Group. The SCD-Well randomized controlled trial: Effects of a mindfulness-based intervention versus health education on mental health in patients with subjective cognitive decline (SCD). Alzheimers Dement (N Y). 2018 Dec 14;4:737-745. doi: 10.1016/j.trci.2018.10.010. eCollection 2018. PMID 30581979
- [Result] Marchant NL, Barnhofer T, Coueron R, Wirth M, Lutz A, Arenaza-Urquijo EM, Collette F, Poisnel G, Demnitz-King H, Schild AK, Coll-Padros N, Delphin-Combe F, Whitfield T, Schlosser M, Gonneaud J, Asselineau J, Walker Z, Krolak-Salmon P, Molinuevo JL, Frison E, Chetelat G, Jessen F, Klimecki OM; The Medit-Ageing Research Group. Effects of a Mindfulness-Based Intervention versus Health Self-Management on Subclinical Anxiety in Older Adults with Subjective Cognitive Decline: The SCD-Well Randomized Superiority Trial. Psychother Psychosom. 2021;90(5):341-350. doi: 10.1159/000515669. Epub 2021 Apr 19. PMID 33873195
- [Result] Whitfield T, Demnitz-King H, Schlosser M, Barnhofer T, Frison E, Coll-Padros N, Dautricourt S, Requier F, Delarue M, Gonneaud J, Klimecki OM, Lutz A, Paly L, Salmon E, Schild AK, Walker Z, Jessen F, Chetelat G, Collette F, Wirth M, Marchant NL; Medit-Ageing Research Group. Effects of a mindfulness-based versus a health self-management intervention on objective cognitive performance in older adults with subjective cognitive decline (SCD): a secondary analysis of the SCD-Well randomized controlled trial. Alzheimers Res Ther. 2022 Sep 6;14(1):125. doi: 10.1186/s13195-022-01057-w. PMID 36068621
- [Result] Schlosser M, Demnitz-King H, Barnhofer T, Collette F, Gonneaud J, Chetelat G, Jessen F, Kliegel M, Klimecki OM, Lutz A, Marchant NL; Medit-Ageing Research Group. Effects of a mindfulness-based intervention and a health self-management programme on psychological well-being in older adults with subjective cognitive decline: Secondary analyses from the SCD-Well randomised clinical trial. PLoS One. 2023 Dec 15;18(12):e0295175. doi: 10.1371/journal.pone.0295175. eCollection 2023. PMID 38100477
- [Result] Demnitz-King H, Gonneaud J, Klimecki OM, Chocat A, Collette F, Dautricourt S, Jessen F, Krolak-Salmon P, Lutz A, Morse RM, Molinuevo JL, Poisnel G, Touron E, Wirth M, Walker Z, Chetelat G, Marchant NL; Medit-Ageing Research Group. Association of Self-reflection With Cognition and Brain Health in Cognitively Unimpaired Older Adults. Neurology. 2022 Sep 27;99(13):e1422-e1431. doi: 10.1212/WNL.0000000000200951. Epub 2022 Jul 19. PMID 35853750